CLINICAL TRIAL: NCT04907864
Title: Effect of Multi-modal Intervention Care on Cachexia in Patients With Advanced Cancer Compared to Conventional Management (MIRACLE): An Open-label, Phase 2 Tria
Brief Title: Effect of Multi-modal Intervention Care on Cachexia in Patients With Advanced Cancer Compared to Conventional Management (MIRACLE)
Acronym: MIRACLE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kil Yeon Lee (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Sponsor-Investigator, Kil Yeon Lee, Professor, Kyunghee University Medical Center
Organization: Kyunghee University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KHMC-HUMANITAS-01
Record Dates: First submitted 2021-05-25; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Gastric Cancer; Colorectal Cancer; Pancreatic Cancer; Biliary Tract Cancer; Lung Cancer; Precachexia; Cachexia
Keywords: cachexia; chemotherapy; cancer; multi-modal intervention; NSAID
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Biliary Tract Neoplasms; Lung Neoplasms; Cachexia; Neoplasms | interventions — Ibuprofen; Omacor

STUDY DESIGN:
Intervention Model Description: An open-label, randomized phase 2 trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIC (Experimental): Multi-modal intervention
  Interventions: Combination Product: Multi-modal intervention
- CPC (No Intervention): Conventional Palliative Care

INTERVENTIONS:
Combination Product: Multi-modal intervention — Daily oral medications: ibuprofen 400 mg three times a day, omega-3-fatty acid 1 g twice a day, Bojungikki-tang 3.75g twice a day, oral nutritional supplement (HAMONILAN SOLN) 200 ml twice a day Weekly physical exercise by physiatrist (60 minutes per visit) Biweekly psychiatric intervention Nutritional counselling total four times during the study period
  Other Names: ibuprofen (Brufen); omega-3-fattyacid (Omacor); Bojungikki-tang (Kracie Bojungikgitang Extract Fine Granule); oral nutritionalsupplement (HARMONILAN SOLN)
  Arms: MIC

SUMMARY:
Background

Cancer Cachexia (CC) is a multi-factorial process characterized by progressive weight loss, muscle mass and fat tissue wasting, and adversely affecting their quality of life and survival in patients with advanced stage of cancer.

Megestrol acetate (MA), which can help maintain body weight in advanced cancer patients, has not been proven to be effective in improving quality of life or lean body mass. Furthermore, its use is often limited due to various adverse event such as Cushing syndrome, adrenal insufficiency, or thromboembolic risk.

CC has a complex and multi-factorial pathophysiology, and there is no established standard treatment.

Hypothesis CC is irreversible once it occurs and is also difficult to suppress its progression with any single treatment modality.

The investigators hypothesized that a multi-modal intervention comprised of anti-inflammation, omega-3-fatty acids, oral nutritional supplement with counselling by nutritionist, physical exercise, psychiatric intervention as well as Bojungikki-tang which mediates immune-modulation and reverse both of chronic inflammation and wasting condition as a complementary and alternative medicine (CAM) could prevent the development of CC or improve the CC in advanced cancer patients during chemotherapy compared to those who received usual supportive.

DETAILED DESCRIPTION:
[PICOT] Population: Patients with recurrent or metastatic solid cancer (gastric, colorectal, pancreas, biliary tract and lung)

Intervention: Multimodal treatment

Comparison: Conventional palliative care

Outcome: Change of total lean body mass, Change of handgrip strength Time: 12 weeks of study period for each subject during the first- or second-line palliative chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients over 19 years of age
* Patients diagnosed with gastrointestinal (stomach, esophageal, direct colon, liver, pancreatic biliary tract) cancer and lung cancer
* Patients receiving first- or second-line palliative chemotherapy
* ECOG PS 0-2
* Patients who were classified as normal, precachexia or cachexia according to the cachexia classification criteria

  * Normal: Neither pre-cachexia Nor cachexia
  * Precachexia: Weight loss ≤5%, Anorexia or glucose intolerance in last 6 months
  * Cachexia: Weight loss >5%, or BMI <20 with weight loss >2% in last 6 months
* Adequate organ functions

Exclusion Criteria:

* Patients with history of heart failure or currently being treated for heart failure
* Patients with SBP of 160 mmHg or higher or DBP of 100 mmHg or higher despite antihypertensive medication
* Patients with or have a history of bronchial asthma
* Patients with bowel obstruction
* Patients who have taken appetite stimulants or anabolic or anti-catabolic agents (eg. Megestrol acetate, progestational agents, etc.) within 30 days prior to the study enrollment
* Patients who received steroid treatment (> 10 mg/d prednisolone or equivalent) within 3 months prior to the study enrollment
* Patients who have taken nonsteroidal anti-inflammatory drugs or aspirin continuously for more than 1 week
* Patients with problems with taking non-steroidal anti-inflammatory drugs (NSAIDs) or those with uncontrolled diabetes due to digestive system diseases (gastric ulcer, gastrointestinal bleeding, etc.)
* Patients who are pregnant or breastfeeding, who have not used proper contraception (oral, injection, infusion or hormonal contraceptive methods, intrauterine devices and blocking methods)
* Patients who are taking anticoagulants (e.g. warfarin or heparin)
* Patients who have difficulty in oral administration
* Patients who have a history of hypersensitivity reactions such as asthma, hives, or allergic reactions to drugs containing ibuprofen, aspirin, and other nonsteroidal anti-inflammatory drugs (including COX-2 inhibitors)
* Patients who showed clinically significant hypersensitivity reactions to investigational products

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Median change (kilogram, kg) in total lean body mass (LBM) | Change of value between baseline and week13
  The average of the change (kg) from baseline at week 7 and change from baseline at week 13 measured by DEXA (dual-energy X-ray absorptiometry)
Median change (kg) in handgrip strength | Change of value between baseline and week13
  The average of the change (kg) from baseline at week 7 and change from baseline at week 13 measured by DEXA (dual-energy X-ray absorptiometry)

SECONDARY OUTCOMES:
Median change (kg) in fat mass | Change of value between baseline and week13
  The average of the change (kg) from baseline at week 7 and change from baseline at week 13 measured by DEXA (dual-energy X-ray absorptiometry)
Median change (kg) in total body mass | Change of value between baseline and week13
  The average of the change (kg) from baseline at week 7 and change from baseline at week 13 measured by DEXA (dual-energy X-ray absorptiometry)
Median change (kg) in body weight (kg) | Change of value between baseline and week13
  The average of the change (kg) from baseline at week 7 and change from baseline at week 13 measured by the calibrated scale
Median change (kg) in lean body mass of trunk | Change of value between baseline and week13
  The average of the change (kg) from baseline at week 7 and change from baseline at week 13 measured by DEXA (dual-energy X-ray absorptiometry)
Median change (kg) in lean body mass of both upper and lower extremities | Change of value between baseline and week13
  The average of the change (kg) from baseline at week 7 and change from baseline at week 13 measured by DEXA (dual-energy X-ray absorptiometry)
Change from Anorexia-Cachexia scale | Change of value between baseline and week 13
  Functional Assessment of Anorexia/Cachexia Treatment (FAACT) version 4, The higher the score, the better the quality of life (QoL) with range 0-156.
Change in quality of life (QoL) | Change of value between baseline and week 13
  The EORTC QLQ-C30 (Version 3) uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
  The EORTC QLQ-C30 (Version 3) uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.
Rate of toxicity with clinical significance, and possible relationship to either study intervention | Change of value between baseline and week 13
  Assessed by the investigator, based on toxicity grade (according to the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Kil Yeon Lee, M.D., Principal Investigator — Kyung Hee University Hospital
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After anonymizing the patient's confidential information, it can be converted into data and shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Maeng CH, Kim BH, Chon J, Kang WS, Kang K, Woo M, Hong IK, Lee J, Lee KY. Effect of multimodal intervention care on cachexia in patients with advanced cancer compared to conventional management (MIRACLE): an open-label, parallel, randomized, phase 2 trial. Trials. 2022 Apr 11;23(1):281. doi: 10.1186/s13063-022-06221-z. PMID 35410294